CLINICAL TRIAL: NCT03083080
Title: Ultrasound-guided Peripheral Nerve Block for Non-intubated Uniportal Video-assisted Thoracoscopic Surgery
Brief Title: VATS Block for Uniportal Video-assisted Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201504056
Record Dates: First submitted 2017-02-20; First posted 2017-03-17 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Efficacy and Safety of VATS Block
MeSH Terms: interventions — Thoracic Surgery, Video-Assisted; Ropivacaine; Epinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VATS block (ropivacaine + epinephrine) (Experimental): VATS block is the peripheral nerve block for video-assisted thoracic surgery, whose injection is administered at the site of chest wall incision.
  Interventions: Procedure: VATS; Drug: Ropivacaine; Drug: Epinephrine

INTERVENTIONS:
Procedure: VATS — VATS is the abbreviation of video-assisted thoracic surgery, which aims to minimize the wound for thoracic surgery and to enhance patient recovery after surgery
Drug: Ropivacaine — 30 mL 0.5% ropivacaine is used to achieve VATS block
Drug: Epinephrine — 1:400000 epinephrine is mixed with ropivacaine (local anesthetic) to reduce the risk of local anesthetic systemic toxicity

SUMMARY:
Traditionally, video-assisted thoracic surgery is performed under general anesthesia with double-lumen endotracheal tube. However, the complications associated with this large tube as well as inhalation anesthetics are frequently reported. Therefore, currently there is a trend toward non-intubated anesthesia methods for video-assisted thoracic surgery, which includes thoracic epidural block, peripheral nerve block, local anesthesia, local combined with peripheral nerve block, etc. Thoracic epidural block demands a high technique, but still risks catastrophic neurological complications in case of accidental dural puncture. Local anesthesia, perhaps more straightforward, however may need supplemental analgesia during incision, which will inevitably interrupt surgery and negatively affect the patients. This study aims to apply ultrasound guidance during local anesthetic injection for local anesthesia-based video assisted thoracic surgery, which helps inject the local anesthetic into the key intercostal nerve plane to provide more specific and precise blockade, thus avoiding the chance of blind injection. At the same time, ultrasound guidance has the potential to reduce the risk of systemic toxicity, prolong the duration of analgesia postoperatively, and facilitates postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adults younger than 80 years old and weighing between 50-90 kg are scheduled for one-port video assisted thoracic surgery .

Exclusion Criteria:

* Anticipated difficult airway
* Obvious coagulation abnormality
* Psychiatric patients or drug addiction
* Emergency operation or patients with a full stomach
* Difficulty in language expression
* Allergic to local anesthetic, morphine, or NSAID
* BMI > 35
* Pregnancy
* Respiratory insufficiency
* Severe pleural adhesion
* Need for pleurodesis
* Refuse patient-controlled analgesia
* Patients with a pacemaker
* Severe liver dysfunction (serum albumin<25g/l or Child-Pugh score≧10)
* Severe kidney dysfunction (creatinine clearance<30ml/min)
* Inflammatory bowel disease
* Congestive heart failure (NYHA II-IV)
* Confirmed ischemic heart disease, peripheral arterial disease and/or cerebral vascular disease
* Patients with a high intra-ocular pressure (e.g. glaucoma)
* Neurological symptoms over the ipsilateral upper part of the body

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-27 (Estimated); Primary Completion 2019-03-26 (Estimated); Study Completion 2019-03-26 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale intraoperatively | During chest wall incision
  Self-reporting pain intensity, pain site, and analgesic dosage during surgery
TIme to lose skin sensation (light touch and thermal) over the injection site | Up to 30 mins after ropivacaine injection
  Skin sensation will be tested every 5 minutes after ropivacaine injection until loss of both sensation (readiness for skin incision)

SECONDARY OUTCOMES:
Ropivacaine concentration at different time points after injection | Up to 120 mins following injection
  Blood sampling at seven time points (10, 20, 30, 45, 60, 90, 120 minutes following injection)
Common characteristics of ultrasound anatomy by analyzing video clips | Three time points (upon obtaining informed consent, prior to injection and during injection)
  Recording the ultrasound images at three time points
Numerical rating scale postoperatively | Up to 72 hours following surgery
  Pain scores evaluated at six time points (at the conclusion of surgery, and at 2h, 6h, 24h, 48h, and 72h post-surgery)